CLINICAL TRIAL: NCT03942354
Title: Patient-reported Experiences and Quality of Life Outcomes in the TB-PRACTECAL Clinical Trial
Acronym: PRACTECAL-PRO
Status: Completed | Type: Observational
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: University of Sussex (Other); London School of Hygiene and Tropical Medicine (Other); THINK TB & HIV Investigative Network (Network); Wits Health Consortium (Pty) Ltd (Other); Ministry of Public Health, Republic of Belarus (Other Government); Ministry of Health, Republic of Uzbekistan (Other Government)
Responsible Party: Sponsor
Other Study IDs: PRACTECAL-PRO
Record Dates: First submitted 2019-02-22; First posted 2019-05-08 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Quality of life, drug-resistant tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — bedaquiline; pretomanid; Moxifloxacin; Linezolid; Clofazimine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention arm: A total of 54 intervention arm trial patients (from TB-PRACTECAL trial) are anticipated across all three sites: South Africa, Belarus, and Karakalpakstan.
  54 matched healthy controls are anticipated.
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Moxifloxacin; Drug: Linezolid; Drug: Clofazimine
- Standard therapy: 54 standard therapy trial patients (from TB-PRACTECAL trial) will be recruited across all three sites. Patients will complete measures at baseline, 3 months, 6 months and 12 months.
  54 matched healthy controls are anticipated.
  Interventions: Drug: Directly observed therapy (DOT)

INTERVENTIONS:
Drug: Bedaquiline — Bedaquiline is a diarylquinoline class antimicrobial which blocks the proton pump for ATP synthase of mycobacteria. This in turn blocks the ATP production required for cellular energy production and leading to cell death.
  Other Names: Sirturo; R207910; TMC207
  Groups: Intervention arm
Drug: Pretomanid — Pretomanid is a nitroimidazole class antimicrobial which interferes with cell wall biosynthesis in mycobacteria. It may have other mechanisms of action as well in non-replicating mycobacteria.
  Other Names: PA-824
  Groups: Intervention arm
Drug: Moxifloxacin — Moxifloxacin is an 8-methoxyquinolone class antimicrobial that is a potent inhibitor of DNA gyrase and topoisomerase IV in bacteria
  Other Names: Avelox, BAY 12-8039
  Groups: Intervention arm
Drug: Linezolid — Linezolid, an oxazolidinone class antimicrobial which works by inhibiting ribosomal protein synthesis. It is approved for Gram-positive bacterial infections, and is increasingly being used for drug resistant TB disease.
  Other Names: Zyvox
  Groups: Intervention arm
Drug: Clofazimine — Clofazimine is a lipophilic riminophenazine licensed for treatment of leprosy. Its mechanism(s) of action remains unclear, but existing evidence suggests production of reactive oxygen species within Mycobacterium tuberculosis is one mechanism.
  Other Names: Lamprene
  Groups: Intervention arm
Drug: Directly observed therapy (DOT) — Standard therapy
  Groups: Standard therapy

SUMMARY:
PRACTECAL-PRO is a sub-study of a TB-PRACTECAL clinical trial for multidrug resistant Tuberculosis. It evaluates the effectiveness of TB-PRACTECAL interventions from the patient perspective in terms of their quality of life, shared decision making and satisfaction with services.

DETAILED DESCRIPTION:
Tolerability of drugs for TB is a complex and dynamic course for patients with drug resistance and can be affected by many different factors. A deeper understanding of the perspectives and experience of men and women participating in novel TB treatment trials will add to the understanding of the safety and efficacy of treatment.

TB-PRACTECAL is a multicentre, open label, phase 2-3 randomised controlled trial evaluating exclusively oral 6 months regimens containing bedaquiline, pretomanid, linezolid +/- moxifloxacin or clofazimine for the treatment of microbiologically confirmed pulmonary M/XDR-TB. It is registered with the ClinicalTrials.gov with identifier number NCT02589782. The trial aims to recruit 630 adults from two sites in Uzbekistan (Nukus and Tashkent) and one site each from Belarus and South Africa.

The TB-PRACTECAL trial assumes that even if the investigational arms would have non-inferior efficacy and safety compared to the standard of care outcomes, patients would prefer a shorter, exclusively oral regimen with a lower pill count. This study therefore aims to describe patient experiences (i.e. the quality of the treatment experience as opposed to the quantity of treatment or the amount of time spent on it).

The PRACTECAL-PRO sub-study aims to answer the question: "What are the perceptions, expectations and experiences of novel TB treatment for adult patients participating in a six-month regimen clinical trial in Uzbekistan, South Africa and Belarus?"

The objectives for the analysis are:

* To compare baseline scores between trial patients (all interventional arm patients plus standard of care patients) with healthy controls.
* To assess changes in scores over time in patients on the intervention arms and patients on the standard of care arm.
* To assess the utility of the SF 12 and SGRQ in a TB clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited into the TB-PRACTECAL trial in the approved sites OR
* Local healthy-controls of a similar profile in terms of age and gender aged ≥18 years AND
* Literate in the study questionnaire languages
* Able to sign the sub-study informed consent form after agreeing to the additional interviews and completion of questionnaires.

Exclusion Criteria:

* TB patients excluded from TB-PRACTECAL clinical trial
* Healthy volenteers with co-morbidities
* Healthy volenteers found to have TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an observational sub-study of parent RCT TB-PRACTECAL (NCT02589782. Arms 1 & are the study population, and a sub-set of the main RCT cohort.
  Local healthy-controls of a similar profile in terms of age and gender aged ≥18 years are also included.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Change in St George's respiratory questionnaire SGRQ survey questionnaire from baseline to 12 months | 12 months
  To assess the quality of life (QoL) of trial patients from baseline to 12 months: both those treated in the investigational arms and the standard of care arm. For the SGRQ, a change of 4 points is suggested to indicate a clinically significant change, although the questionnaire was developed with patients who had COPD rather than TB. In the sub-study with a relatively small sample we cannot be confident about whether a change of 4 points represents a similarly significant change, but we will be mindful to assess this possibility. Ultimate aim is to determine whether disease-specific patient quality of life scores improve in investigational arm patients from baseline to successful completion of treatment.
Changes in Short form 12 survey questionnaire (patient satisfaction and experience) from baseline to 12 months | 12 months
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). Ultimate aim is to determine whether disease-specific patient satisfaction scores improve in investigational arm patients from baseline to successful completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Beverley Stringer, Principal Investigator — MSF
Locations (6):
- Republican Scientific and Practical Centre for Pulmonology and Tuberculosis hospital, Minsk, Belarus
- South Africa (3):
  - THINK Clinical Trial Unit, Hillcrest, Durban, KwaZulu-Natal
  - Doris Goodwin Hospital, Pietermaritzburg, KwaZulu-Natal
  - Helen Jospeh Hospital, Johannesburg
- Uzbekistan (2):
  - Republican TB Hospital No. 2, Nukus, Karakalpakstan
  - Sh Alimov Republican Specialised Scientific-Practical Medical Centre for Phthysiology and Pulmonology Hospital, Tashkent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stringer B, Lowton K, James N, Nyang'wa BT. Capturing patient-reported and quality of life outcomes with use of shorter regimens for drug-resistant tuberculosis: mixed-methods substudy protocol, TB PRACTECAL-PRO. BMJ Open. 2021 Sep 6;11(9):e043954. doi: 10.1136/bmjopen-2020-043954. PMID 34489263